CLINICAL TRIAL: NCT00535015
Title: A Randomized, Double-Blind, Pilot Study Comparing the Safety and Efficacy of Betamarc Plus Chemotherapy to Chemotherapy Alone in the Prevention and Treatment of CACS in Patients With Advanced NSCLC
Brief Title: Safety and Efficacy Study of Betamarc to Treat Loss of Weight and Appetite in Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Objectives of study could not be met within a reasonable timeframe.
Sponsor: Anaborex (Industry)
Responsible Party: Jeff Rudy, Vice President Clinical Operations, Anaborex, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANA-CTP0002
Record Dates: First submitted 2007-09-23; First posted 2007-09-26 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Anorexia; Cachexia; Weight Loss; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Anorexia; Cachexia; Weight Loss; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Betamarc — 2 tabs BID

SUMMARY:
The purpose of this study is to determine whether Betamarc is effective in improving the appetite and reversing weight loss in patients with advanced Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stage IIIB or IV non-resectable NSCLC. Recurrent disease after resection for earlier stage disease is acceptable as long as patients are at least 6 months from surgery.
* Treatment plan includes a platinum-based doublet chemotherapy.
* ECOG 0, 1 or 2.
* Self-reported loss of body weight or anorexia.
* Serum C-reactive protein ≥5 mg/L.
* Life expectancy of at least 6 months.
* Adequate bone marrow, liver and renal function.
* Normal serum potassium.
* Ability to comply with the study requirements and give written informed consent.

Exclusion Criteria:

* Known physical or functional obstruction of the gastrointestinal tract, malabsorption, intractable vomiting, uncontrollable diarrhea, concurrently receiving tube feeding or parenteral nutrition, or unable to swallow investigational drug product.
* Concomitant therapy with an appetite stimulant.
* History of poorly controlled hypertension or congestive heart failure.
* Any implanted devices that could interfere with DXA scanning.
* Prolongation of QT interval.
* History of additional risk factors for torsades de pointe.
* Concomitant therapy with beta-adrenergic receptor antagonists (beta-blockers) or ergot derivatives.
* Females who are breast feeding, pregnant or of child-bearing potential who are not using adequate birth control.
* Any second malignancy which might confound the interpretation of safety or efficacy assessments.
* Any condition which increases the patient's risk for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Functional capacity (strength and endurance), body composition by DXA, inflammation, patient reported outcomes, anti-tumor response rate | 25 weeks

SECONDARY OUTCOMES:
Adverse events, ECG, vital signs, clinical laboratory parameters and physical examination | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yung-chuan Sung, Principal Investigator — Cathay General Hospital; Hsing-jin Eugene Liu, Principal Investigator — Taipei Medical University Muncipal Wan Fang Hospital; Te-chun Hsia, Principal Investigator — China Medical University Hospital; Gee-chen Chang, Principal Investigator — Taichung Veterans General Hospital; Yao-kuang Wu, Principal Investigator — Tzu Chi General Hospital Taipei Branch; Kwok-keung Yuen, Principal Investigator — Tuen Mun Hospital; Daniel Chua, Principal Investigator — Queen Mary Hospital, Hong Kong; Chung-kong Kwan, Principal Investigator — The Queen Elizabeth Hospital; Kwok-chi Lam, Principal Investigator — Prince of Wales Hospital; Dae-ho Lee, Principal Investigator — Asan Medical Center; Jong-seok Lee, Principal Investigator — Seoul National University Bundang Hosptial; Hoon-kyo Kim, Principal Investigator — Saint Vincent's Hospital, Korea; Jin-hyoung Kang, Principal Investigator — The Catholic University of Korea, St. Mary's Hospital; Anita Zarina binti Bustam, Principal Investigator — University of Malaya; Abdul Razak bin Abdul Muttalif, Principal Investigator — Penang Hospital, Malaysia; Biswa Mohan Biswal, Principal Investigator — Hospital Universiti Sains Malaysia; Wu-chou Su, Principal Investigator — National Cheng-Kung University Hospital; Ming-lin Ho, Principal Investigator — Chunghua Christian Hospital; Chang-yao Tsao, Principal Investigator — Chung Shan Medical University; Cheng-ta Yang, Principal Investigator — Chang Gung Memorial Hospital, Chiayi; Wen-Tsung Huang, Principal Investigator — Chi Mei Medical Center Liou-Ying Campus; Edy Suratman, Principal Investigator — Dharmais Cancer Hospital; Elisna Syahruddin, Principal Investigator — Persahabatan Hospital; Alexander Ginting, Principal Investigator — Gatot Subroto Central Army Hospital
Locations (6):
- China (2):
  - Queen Elizabeth Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Cathay General Hospital, Taipei
  - Taipei Medical University Muncipal Wan Fang Hospital, Taipei